CLINICAL TRIAL: NCT07202364
Title: A Multicenter, Open-Label, Phase II Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of YL202 in Selected Patients With Advanced Solid Tumors
Brief Title: A Study of YL202 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL202-CN-203-01
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer; Colorectal Cancer; Cervical Cancer; Locally Advanced or Metastatic Solid Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A, B, D and E (Experimental): This includes a dose-exploration period and a dose-expansion period.
  Interventions: Drug: YL202
- Cohort C (Experimental): This includes a dose-exploration period and a dose-expansion period. Participants in Cohort C will be randomized in a 1:1 ratio to one of the two dose levels.
  Interventions: Drug: YL202

INTERVENTIONS:
Drug: YL202 — YL202 will be intravenously infused over 60±10 min

SUMMARY:
This study is a multicenter, open-label, phase II study of YL202 in China to evaluate the efficacy, safety, and PK characteristics of YL202 in selected patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, phase II study of YL202 in China to evaluate the efficacy, safety, and PK characteristics of YL202 in the advanced non small cell lung cancer/colorectal cancer/cervical cancer, etc. YL202 is an antibody-drug conjugate (ADC) that targets HER3 protein

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following criteria to be included in the study:

  1. Subjects who are aware of relevant study information prior to the start of the study, and voluntarily sign and date on the informed consent form (ICF).
  2. Subjects aged ≥18 years at the time of giving informed consent
  3. Body mass index (BMI) within the range of 18 to 32 kg/m2.
  4. Subjects with histologically or cytologically confirmed non-Sq NSCLC/CRC/CC or other advanced solid tumor, and had received 1-2 lines of systemic therapy in the advanced/metastatic setting
  5. There is at least one extracranial measurable lesion as the target lesion per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
  6. Archived or fresh tumor tissue samples are available.
  7. Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
  8. The function of organs and bone marrow meets the requirements within 7 days prior to the first dose
  9. Female subjects of childbearing potential must agree to adopt highly effective contraceptive measures from screening throughout the study period and within at least 6 months after the last dose of the investigational product. Male subjects must agree to adopt highly effective contraceptive measures from screening throughout the study period and within at least 6 months after the last dose of the investigational product.
  10. Expected survival ≥3 months.
  11. Be capable of and willing to comply with the visits and procedures stipulated in the study protocol.

Exclusion criteria

* Subjects who meet any of the following criteria should be excluded from the study:

  1. Prior drug therapy targeting HER3
  2. Previously intolerant to topoisomerase I inhibitors or ADC therapy composed of topoisomerase I inhibitors).
  3. Are participating in another clinical study, unless it is an observational (non-interventional) clinical study or in the follow-up period of an interventional study.
  4. The washout period from the previous anti-tumor therapy is insufficient prior to the first dose of the investigational product.
  5. Patients who received major surgery (excluding diagnostic surgery) within 4 weeks prior to the first dose of the investigational product or those who are expected to receive major surgery during the study.
  6. Prior treatment with allogeneic bone marrow transplantation or solid organ transplantation.
  7. Prior treatment with systemic steroids (prednisone >10 mg/day or equivalent) or other immunosuppressive treatment within 2 weeks prior to the first dose of the investigational product.
  8. Patients who received any live vaccine within 4 weeks prior to the first dose of the investigational product or those who plan to receive live vaccine during the study period.
  9. Meningeal metastasis or cancerous meningitis.
  10. Brain metastasis or spinal cord compression.
  11. Patients with uncontrolled or clinically significant cardiovascular diseases.
  12. Clinically significant complicated pulmonary disorders.
  13. Medical history of hepatic encephalopathy within 6 months prior to the first dose.
  14. Subjects with active or chronic corneal disorders, or other active eye disorders requiring continuous treatment, or any clinically significant corneal disorders that preclude adequate monitoring of drug-induced keratopathy.
  15. Diagnosed with Gilbert's syndrome.
  16. Significantly symptomatic or unstable pleural effusion, peritoneal effusion, and pericardial effusion, or those requiring repeated drainage.
  17. Medical history of gastrointestinal perforation and/or fistula within 6 months prior to the first dose, or active gastric and duodenal ulcers, ulcerative colitis, or other gastrointestinal diseases that may cause hemorrhage or perforation in the opinion of the investigator.
  18. Serious infection prior to the first dose (National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0 grade ≥3),
  19. Patients with severe coagulopathy or other diseases with evident risk of bleeding.
  20. Patients with uncontrolled diabetes mellitus.
  21. Human immunodeficiency virus (HIV) infection; positive syphilis antibody and a positive titer result.
  22. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
  23. Medical history of any other primary malignancies within 5 years prior to the first dose of the investigational product, except fully resected non-melanoma skin cancer, cured in-situ disease, or other cured solid tumors.
  24. Unresolved toxicity of previous anti-tumor therapy,
  25. History of severe hypersensitivity to inactive ingredients in the drug substance (DS) and drug product (DP) or other monoclonal antibodies.
  26. Lactating women, or women who are confirmed pregnant via a pregnancy test within 3 days prior to the first dose.
  27. Have any diseases, medical conditions, organ system dysfunction, or social conditions that may interfere with the subject ability to sign the ICF, adversely affect the subject ability to cooperate and participate in the study, or affect the interpretation of study results, including but not limited to mental illness or substance/alcohol abuse, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 3 years
  ORR: defined as the proportion of patients who achieved a best overall response of complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 3 years
  PFS: defined as the time interval from the date of the first dose of study drug to the date of first documentation of PD or death due to any cause, whichever occurs first.
Depth of response (DpR) | Up to approximately 3 years
  DpR: defined as the proportion of target lesion shrinkage from baseline to maximum tumor size.
Disease control rate (DCR) | Up to approximately 3 years
  DCR: defined as the proportion of patients who achieved a best overall response of complete response (CR), partial response (PR) or stable disease (SD).
Duration of response (DoR) | Up to approximately 3 years
  DoR: defined as the time interval from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progressive disease (PD).
Time to response (TTR) | Up to approximately 3 years
  TTR: defined as the time interval from the date of the first dose of study drug to the date of the first documentation of objective response (CR or PR).
Overall survival (OS) | Up to approximately 3 years
  OS: defined as the time interval from the date of the first dose of study drug to the date of death due to any cause.
Nature and frequency of adverse events (AEs) with severity | Up to approximately 3 years
  Nature and frequency of AEs with severity is aim to evaluate the safety of YL202.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Tumor Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No